CLINICAL TRIAL: NCT00633919
Title: A Randomised, Double-blind, Placebo-controlled Trial Assessing the Efficacy of SLITone in House Dust Mite Allergic Patients
Brief Title: Efficacy of SLITone in House Dust Mite Allergic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Santiago Martín -Trial Manager; ALK-Abelló S.A., ALK-Abelló S.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E02/04/SLIT1-M; EudraCT - 2005-004731-21
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Allergy
Keywords: House dust mites; Sublingual immunotherapy; Allergy; Allergic asthma
MeSH Terms: conditions — Hypersensitivity | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Prednisone; desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): SLITone Dermatophagoides Mix
  Interventions: Biological: SLITone(TM) Dermatophagoides mix; Drug: Salbutamol inhaler; Drug: Budesonide/formoterol inhaler; Drug: Prednisone tablet; Drug: Desloratadine tablet; Drug: Budesonide nasal spray
- Placebo (Placebo Comparator): SLITone Placebo
  Interventions: Biological: Placebo; Drug: Salbutamol inhaler; Drug: Budesonide/formoterol inhaler; Drug: Prednisone tablet; Drug: Desloratadine tablet; Drug: Budesonide nasal spray

INTERVENTIONS:
Biological: SLITone(TM) Dermatophagoides mix — Sublingual immunotherapy with SLITone Dermatophagoides mix (200 STU) once daily for 2 years
  Arms: Active
Biological: Placebo — Sublingual immunotherapy once daily for 2 years
  Arms: Placebo
Drug: Salbutamol inhaler — 200 µg per puff; a short acting beta2-agonist (please refer to the 'detailed description' for details on the use)
  Other Names: Ventilastin
Drug: Budesonide/formoterol inhaler — 80/4.5 µg per inhalation; a combination of inhaled corticosteroids and long acting beta2-agonist (please refer to the 'detailed description' for details on the use)
  Other Names: Symbicort
Drug: Prednisone tablet — 5 mg per tablet; oral corticosteroids (please refer to the 'detailed description' for details on the use)
Drug: Desloratadine tablet — 5 mg per tablet: anti-histamine (please refer to the 'detailed description' for details on the use)
  Other Names: Aerus
Drug: Budesonide nasal spray — 64 µg per puff; inhaled corticosteroid (please refer to the 'detailed description' for details on the use)

SUMMARY:
This trial has been designed to evaluate the efficacy of specific immunotherapy with SLITone Dermatophagoides mix compared with placebo in subjects with house dust mite allergic asthma, based on asthma medication use during a period of 2 months with a high environmental exposure to mites (autumn 2008).

DETAILED DESCRIPTION:
This trial was conducted as a multi-centre, randomised, double-blind, parallel-group, placebo-controlled phase III trial, assessing the efficacy of SLITone Dermatophagoides mix in adults (18-65 years). 5 centres in Spain participated.

Subjects with house dust mite allergic asthma were randomised to receive either SLITone Dermatophagoides mix (active) or placebo treatment (1:1) for approximately 1 year. The trial duration was extended to 2 years. Administration was done sublingually (under the tongue) once daily preferably in the morning. A monodose container comprised the daily dose of 200 STU.

Subjects were kept in asthma control during the entire trial (2 years). Except for during 2 evaluation periods of 2 months in autumn 2007 and autumn 2008, subjects used the medications prescribed by their physician. During the 2 evaluation periods of 2 months in autumn 2007 and autumn 2008, subjects used provided and standardised rhinoconjunctivitis and asthma medications. The asthma medication use was to reflect the subject's asthma status. This was done by treatment with a low maintenance dose of control medication supplemented with rescue medication as needed.

Rhinoconjunctivitis medication during the 2 evaluation periods in autumn 2007 and autumn 2008; to standardise the medication used to relieve rhinoconjunctivitis symptoms, subjects were provided with the following free medications as needed:

* Desloratadine tablet (5 mg per tablet; anti-histamine; Aerus®)
* Budesonide nasal spray (64 µg per puff; inhaled corticosteroid)
* Prednisone tablet (5 mg per tablet; oral corticosteroid)

Subjects were instructed to use this medication instead of their usual medication during the 2 evaluation periods in autumn 2007 and autumn 2008, and to record the used medication and symptoms in the daily diary.

Asthma medication during the evaluation period in autumn 2007; prior to the 2 months evaluation period in autumn 2007, the asthma control medication use was interrupted to obtain a medication-free period. Subjects were provided with the following free medications to standardise the treatment used to relieve asthma symptoms:

* Salbutamol inhaler (200 µg per puff; a short acting β2-agonist; Ventilastin®).
* Budesonide/formoterol inhaler (80/4.5 µg per inhalation; a combination of inhaled corticosteroids and long acting β2-agonist; Symbicort®).
* Prednisone tablet (5 mg per tablet; oral corticosteroid).

Subjects were instructed to use this medication instead of their usual medication during the evaluation period in autumn 2007 as follows:

They were to use salbutamol inhaler as asthma rescue medication until they either:

* needed more than 4 inhalations of salbutamol per day for 2 consecutive days
* suffered from nocturnal asthma forcing them to wake up
* suffered from exercise-induced dyspnoea doing ordinary tasks In these cases, subjects were to contact the investigator to determine the amount of budesonide/formoterol to use as daily asthma control medication. The budesonide/formoterol inhaler was thereafter to be used as rescue medication as needed instead of salbutamol. Prednisone could be used as a last option.

Asthma medication during the evaluation period in autumn 2008: At the 2 months evaluation period in autumn 2008, subjects were maintained at a low dose of budesonide/formoterol (daily asthma control medication) and they used the budesonide/formoterol inhaler as rescue medication as needed. Prednisone could be used as a last option.

Asthma medication used during the evaluation periods in autumn 2007 and autumn 2008 were recorded in a daily diary.

One primary efficacy endpoint and 16 secondary efficacy endpoints were assessed; the result of the primary efficacy endpoint, 3 secondary endpoints and adverse event reportings are posted here. None of the other secondary endpoints demonstrated a difference between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of house dust mite induced persistent mild to moderate. asthma, with or without concurrent rhinoconjunctivitis, of at least 1 year of evolution.
* Demonstration of a positive specific serum IgE test to Dermatophagoides during the year prior to the screening visit (CAP Class 2 or higher or equivalent).
* Positive Skin Prick Test response (wheal diameter ≥ 3 mm) to Dermatophagoides mix.
* If pre-menopausal female of childbearing potential, the subject must test negative on standard urine pregnancy test.
* Willingness to comply with this protocol.

Exclusion Criteria:

* FEV1 < 70% of predicted value with appropriate medication.
* Asthma controlled at randomization without need of inhaled corticosteroids or with a dose higher than 1000 µg/day of beclometasone or equivalent.
* A clinical history of symptomatic perennial allergic asthma caused by allergens to which the subjects is regularly exposed (Alternaria, cat), other than house dust mites.
* Chronic sinusitis.
* Aspirin or sulfite intolerance.
* Chronic obstructive pulmonary disease.
* Current severe atopic dermatitis.
* Severe asthma.
* Use of an investigational drug within 30 days prior to screening.
* Previous immunotherapy with house dust mite allergens for at least 2 years within the previous 10 years.
* At randomisation, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process (se-rous otitis media is not an exclusion criterion).
* Physical examination with clinically relevant findings.
* Any of the following underlying conditions known or suspected to be present: Cystic fibrosis, malignancy, insulin-dependent diabetes, malabsorption or malnutrition, renal or hepatic insufficiency, chronic infection, drug dependency or alco-holism, ischaemic heart disease or angina requiring current daily medication or with any evidence of disease making implementation of the protocol or interpretation of the protocol results difficult or jeopardising the safety of the subject (e.g. clinically significant cardiovascular, serious immunopathologic, immunodeficiency whether acquired or not, hepatic, neurologic, psychiatric, endocrine, or other ma-jor systemic disease).
* Immunosuppressive treatment.
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the trial, and/or evidence of an uncooperative attitude.
* Unlikely to be able to complete the trial.
* Unwillingness to comply with trial protocol regimen for asthma and/or rhinoconjunctivitis medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Martín, PhD, Study Chair — Clinical Research Director, ALK-Abelló, S.A.
Locations (1):
- Fernando Rodríguez, Santander, Cantabria, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 22 June 2006
Period: Overall Study
Arm/Group | Active | Placebo
Started | 63 | 61
Completed | 36 | 39
Not Completed | 27 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 63 | 61 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 61 | 124
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (8.0) | 30 (9.0) | 31 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  Spain | 63 | 61 | 124

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Asthma Medication Score During a 2-months Evaluation Period in Autumn 2008
Description: Scoring per inhalation/tablet: 1-2 inhalations twice daily of salbutamol (200 ug per inhalation), 2 scores; 1-2 inhalation twice daily of budesonide/formoterol 80 (4.5 ug per inhalation), 4 scores; 1 inhalation twice daily of budesonide/formoterol 160 (4.5 ug per inhalation), 8 scores; up to 10 tablets once daily of prednisone (5 mg), 1.6 scores. The total maximum daily scores were 40.
  The daily score for each medication step was calculated by multiplying the score per inhalation/tablet with the number of inhalations/tablets used (entered as units in the daily diary by the subject).
Time Frame: 8 weeks
Population: Data were based on subjects from the Full Analysis Set (FAS; all randomised subjects following the ITT ICH principle) who had at least one record in the daily diary in the 2 months evaluation period in autumn 2008. All available data were used to their full extent, but no imputation of data was performed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 36 | 39
Scores on a scale | 4.4 (5.9) [2.12 to 6.71] | 4.7 (5.4) [2.45 to 6.88]
Statistical Analysis 1: Comparison: Active vs Placebo; The null hypothesis is the hypothesis of no difference and the alternative to the null hypothesis is the hypothesis of a difference; Test type: Superiority or Other; p = 0.85, Linear mixed effect (LME) model

2. Secondary Outcome: Average Daily Asthma Medication Score During a 2-months Evaluation Period in Autumn 2007
Description: as for outcome 1
Time Frame: 8 weeks
Population: Data were based on subjects from the Full Analysis Set (FAS; all randomised subjects following the ITT ICH principle) who had at least one record in the daily diary in the 2 months evaluation period in autumn 2007. All available data were used to their full extent, but no imputation of data was performed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 48 | 49
Scores on a scale | 4.1 (5.1) | 3.6 (3.9)
Statistical Analysis 1: Comparison: Active vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.52, Linear mixed effect (LME) model

3. Secondary Outcome: Global Evaluation of Efficacy by Subject at the End of The Evaluation Period in 2008
Description: The treatment efficacy was rated by subjects at the end of the evaluation period in autumn 2008. Subjects rated their asthma symptoms in comparison to previous autumn using the categories: "much worse", "worse", "the same", "better", or "much better".
  The categories "much better" or "better" were grouped as "improved". The categories "the same", "worse" or "much worse" were grouped as "not improved".
Time Frame: 8 weeks
Population: All analyses were on all randomised participants (full analysis set) with data in 2008: All available data were used to their full extent, but no imputation of data was performed.
Measure: Number; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 41
Participants
  Subject evaluation: Improved | 28 | 28
  Subject evaluation: Not improved | 8 | 13
  Subject evaluation: Missing data | 1 | 0
Statistical Analysis 1: Comparison: Active vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Proportional odds regression

4. Secondary Outcome: Global Evaluation of Efficacy by Investigator at the End of the Evaluation Period in Autumn 2008
Description: The treatment efficacy was rated by investigators at the end of the evaluation period in autumn 2008. Investigators rated the asthma symptoms in comparison to when subjects entered the trial, using the categories: "much worse", "worse", "the same", "better", or "much better".
  The categories "much better" or "better" were grouped as "improved". The categories "the same", "worse" or "much worse" were grouped as "not improved".
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 41
Participants
  Investigator evaluation: Improved | 30 | 24
  Investigator evaluation: Not improved | 7 | 17
  Investigator evaluation: Missing data | 0 | 0
Statistical Analysis 1: Comparison: Active vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0486, Proportional odds regression

5. Secondary Outcome: Global Evaluation of Efficacy by Subject and Investigator at the End of the Evaluation Period in Autumn 2007
Description: The treatment efficacy was rated by both subject and investigator at the end of the evaluation period in autumn 2007. Subjects rated their asthma symptoms in comparison to previous autumns and investigators rated the asthma symptoms in comparison to when subjects entered the trial, using the categories: "much worse", "worse", "the same", "better", or "much better".
  The categories "much better" or "better" were grouped as "improved". The categories "the same", "worse" or "much worse" were grouped as "not improved".
Time Frame: 8 weeks
Population: All analyses were on all randomised participants (full analysis set) with data in 2007: All available data were used to their full extent, but no imputation of data was performed.
Measure: Number; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 47 | 47
Participants
  Subject evalution: Improved | 30 | 33
  Subject evaluation: Not improved | 17 | 14
  Investigator evaluation: Improved | 33 | 30
  Investigator evaluation: Not improved | 14 | 17
Statistical Analysis 1: Comparison: Active vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Proportional odds regression

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 2/63 | 2/61
Other Adverse Events (participants affected / at risk) | 24/63 | 21/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=63) | Placebo (N=61)
Perianal abscess (Infections and infestations) | 0 (0) | 1 (1) — Unlikely related to specific immunotherapy, moderate in severity
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) — Unlikely related to specific immunotherapy, severe
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unlikely related to specific immunotherapy, severe
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unlikely related to specific immunotherapy, severe
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=63) | Placebo (N=61)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 13 (16) | 9 (10)
Nasopharyngitis (Infections and infestations) | 9 (17) | 14 (18)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Retrospectively, trial design (medication use did not reflect the asthma status of subjects), and subject number (low power) and characteristics (mild, well-controlled asthma; low medication use needed) were not optimal for this trial purpose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ALK must receive copies of any intended communication in advance of publication (at least 15 working days for an abstract or oral presentation and 45 working days for a journal submission). ALK will review the communications for accuracy (thus avoiding potential discrepancies with submissions to health authorities), verify that confidential information is not being inadvertently divulged and provide any relevant supplementary information.